CLINICAL TRIAL: NCT05044728
Title: The Exploration of Immunodynamic Monitoring in the Population Evaluation of Neoadjuvant Chemotherapy Immunotherapy in Patients With Solid Tumor of the Chest.
Brief Title: Exploration of Immunodynamic Monitoring in the Population Evaluation of Neoadjuvant Chemotherapy Immunotherapy in Patients With Solid Tumors of the Chest.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sichuan Cancer Hospital and Research Institute (Other)
Responsible Party: Principal Investigator, Qiang Fang,MD, Principal Investigator, Clinical Professor., Sichuan Cancer Hospital and Research Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTIO1.0
Record Dates: First submitted 2021-09-03; First posted 2021-09-16 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Non-small Cell Lung Cancer; Esophageal Squamous Cell Carcinoma
Keywords: Anti-PD-1; NSCLC; ESCC; Neoadjuvant; Immune microenvironment
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Esophageal Squamous Cell Carcinoma | interventions — Paclitaxel; Carboplatin

STUDY DESIGN:
Intervention Model Description: This study is a prospective, single-arm, open cohort study (randomly stratified within the group).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neoadjuvant Chemotherapy Immunotherapy stage (Experimental): Patients with locally advanced non-small cell lung cancer and locally advanced thoracic esophageal squamous cell carcinoma who met the entry and discharge criteria will be enrolled. After detecting the functional subsets of peripheral CD8-positive T cells, the group was randomly stratified 1:1, respectively. Group A received immunotherapy 24 hours after chemotherapy, and group B received chemotherapy 24 hours after immunotherapy.
  Interventions: Drug: Anti-PD-1 antibody combined with Paclitaxel and carboplatin.; Procedure: Surgical treatment stage

INTERVENTIONS:
Drug: Anti-PD-1 antibody combined with Paclitaxel and carboplatin. — Anti-PD-1 antibody, 240 mg, IV infusion for 30min (not less than 20min and not more than 60min), d1, every 3 weeks for total 2 cycles. Stratified regimen: group A, 24 hours after the end of chemotherapy; Group B will be given immunotherapy on the first day of each cycle.
  Paclitaxel, 135 mg/m2, IV, d1, q3w, for total 2 cycles. Carboplatin, AUC=5 (according to Calvert formula), IV, d1, every 3 weeks for a total of 2 cycles. Stratified regimen: group A, chemotherapy will be given on day 1 of each cycle; Group B will be given chemotherapy drugs 24 hours after the end of immunotherapy.
Procedure: Surgical treatment stage — After the completion of neoadjuvant immunochemotherapy, patients will be tested again for the functional subsets of peripheral CD8 positive T cells. Alternative treatments will be sought for inoperable patients. For patients who are operable will receive minimally invasive or open surgery was performed 1 month after completion of neoadjuvant chemotherapy immunotherapy, and the functional subsets of peripheral CD8 positive T cells were detected again after surgery.

SUMMARY:
Chest malignant solid tumor (mainly lung and esophageal cancer) is a common malignant tumor that seriously threatens the health of residents in China. Its morbidity and mortality rank first, sixth, first, and fourth among all malignant tumors respectively. The treatment effect is not satisfactory, and the overall 5-year survival rate after surgery alone is about 20%-35%. Recent studies have shown that neoadjuvant therapy combined with surgery in the treatment of locally advanced esophageal cancer and lung cancer can significantly improve the efficacy compared with surgery alone. The results of multiple international and multi-center neoadjuvant immunotherapy showed that this new model of combined immunoadjuvant immunotherapy brought a breakthrough point for the treatment of malignant solid tumors of the chest. However, its safety and target benefit groups are still the biggest problems, and there is a large room for improvement. To develop the optimal treatment strategy, it is necessary to further clarify the immunomodulatory mechanisms of neoadjuvant CTIO, explore and develop new evaluation methods and prognostic biomarkers for the selection of targeted benefit patients, and the evaluation of efficacy. This is a key scientific issue in the current neoadjuvant CTIO treatment mode for thoracic malignant solid tumors, mainly lung and esophageal squamous cell carcinoma, which urgently needs to solve its safety and select the benefit population.

DETAILED DESCRIPTION:
As a major participant in cellular immunity, CD8-positive T cells are considered to be the main anti-tumor immune effector cells. In addition to producing specific immune responses to viruses and other infections, their functional subsets are closely related to the occurrence and development of major human diseases. Therefore, we have reason to believe that the combination of dynamic monitoring of host immune background and traditional clinical evaluation can effectively clarify the immune background of patients with lung cancer and esophageal squamous cell carcinoma, and provide new ideas and methods for the selection of appropriate immunotherapy regimen and prognosis evaluation. However, the research in this field is still in its infancy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with locally advanced non-small cell lung cancer (stage II or III) and thoracic esophageal squamous cell carcinoma (CT2N1-2M0, CT3-4AN0-2M0).
* Preoperative biopsy pathology confirmed squamous cell carcinoma or adenocarcinoma with negative driver gene.
* Without any anti-tumor therapy.
* Endoscopic examination indicated that the midpoint of the tumor was located in the middle and lower esophageal thoracic segments.
* Preoperative staging is II or III.
* Ages 18 to 72 years.
* Cardiopulmonary, liver and kidney function tests can tolerate surgery.
* ECOG PS 0-1.
* Signed the informed consent to participate in the study plan before enrollment.

Exclusion Criteria:

* Preoperative endoscopic biopsy pathology confirmed small cell carcinoma.
* Has undergone other anti-tumor therapy.
* Endoscopic examination indicated that the midpoint of the tumor was located in the upper part of the esophagus.
* Preoperative examination suggested that T4B was unresectable or distantly metastatic.
* Corticosteroids or other immunosuppressive drugs were used within 14 days before enrollment. Topical substitute steroids (daily dose ≤10mg) or short-term prescription corticosteroids (≤7 days) were allowed for the prevention or treatment of non-autoimmune diseases.
* A history of active autoimmune disease or a possible recurrence of autoimmune disease.
* Severe chronic or active infectious disease.
* History of interstitial lung disease.

Ages: 18 Years to 72 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-04-01 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Functional subsets of peripheral CD8 positive T cells | Approximately 1 years
Overall response rate(ORR) | Approximately 1 years
  Objective Response Rate is defined as complete response (CR) + partial response (PR), from the beginning of regimental therapy to the end of neoadjuvant therapy, the efficacy of baseline target lesions was assessed by RECIST 1.1 criteria.
Pathological complete response (pCR) | At time of surgery
  Pathological complete response is defined as 0% survival of tumor cells in surgically resected tumor samples after neoadjuvant therapy, as assessed by tumor regression grade.
Immune Related Adverse Events (irAEs) | Approximately 1 years
  Assess all adverse events according to the NCI Common Terminology Criteria for (NCI-CTCAE) v 4.0.3.

SECONDARY OUTCOMES:
Progress Free Survival(PFS) | Approximately 1 years
  Progress Free Survival is defined as included the development of new metastases, or local progression of metastases or primary lesions that underwent surgical resection and will be assessed according to RESIST 1.1 criteria.
2-year survival rate | up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Qiang Fang, PH.D, Principal Investigator — Sichuan Cancer Hospital and Research Institute
Locations (1):
- Sichuan Cancer Hospital, Chengdu, Sichuan, China